CLINICAL TRIAL: NCT03237468
Title: Effectiveness of a Neck Strengthening Program for the Prevention or Mitigation of Sports Concussion Injuries in Student Athletes
Brief Title: Neck Strengthening Program for the Prevention or Mitigation of Sports Concussion
Acronym: PCONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CentraCare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSR#17-4360
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Concussion, Brain
Keywords: concussion; football; student; athlete; sports
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise arm (Experimental): This arm will perform twice weekly neck strengthening exercises.
  Interventions: Other: Neck strengthening exercise to prevent concussion

INTERVENTIONS:
Other: Neck strengthening exercise to prevent concussion — Neck strengthening exercise to prevent concussion in student athletes.

SUMMARY:
Study looks to determine effectiveness of neck strengthening to reduce the incident, duration, and severity of sports related concussion in student athletes.

DETAILED DESCRIPTION:
After recruitment, subjects will have neck strength measured as baseline in addition to doing SCAT5 for baseline and eye tracking, funding pending, in order to compare later assessment for concussion. Throughout study, subject will perform basic, unweighted and weighted neck strengthening exercises twice a week. Periodic re evaluations of neck strength will be performed in order to determine progress. Any time a subject incurs a sports related concussion, a SCAT5 assessment, and eye tracking funding pending, will be done and compared to baseline to measure severity of injury. Weekly follow ups will be done to assess duration of concussion. All measurements, assessments, and exercises are non-invasive and provide minimal risk to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Involved in programmatic athletic activities with an ongoing duration of at least 4 weeks.
* Written informed consent obtained by the subject or subject's legal guardian.
* Written assent from subjects ages 8 years old and above
* Subject is between the ages of 5 and 22 years, male or female.
* Subjects from all racial and ethnic origins will have an opportunity to participate.

Exclusion Criteria:

- Corrected vision less than 20/500.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-08-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Effect of increase in neck strength in reducing risk of concussion | One year
  Neck strength, as measured by a dynamometer, will be assessed and compared to baseline. Magnitude in strength will be analyzed in relation to incidence, severity, and duration of concussion.

SECONDARY OUTCOMES:
Effect of baseline neck strength on risk of concussion | One year
  Risk of concussion will be analyzed in relation to baseline strength measurements to assess overall effect of neck strength.

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Samadani, MD, PhD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Eckner JT, Oh YK, Joshi MS, Richardson JK, Ashton-Miller JA. Effect of neck muscle strength and anticipatory cervical muscle activation on the kinematic response of the head to impulsive loads. Am J Sports Med. 2014 Mar;42(3):566-76. doi: 10.1177/0363546513517869. Epub 2014 Jan 31. PMID 24488820
- [Background] Dugan S, Seymour L, Roesler J, Glover L, Kinde M. This is your brain on sports. Measuring concussions in high school athletes in the Twin Cities metropolitan area. Minn Med. 2014 Sep;97(9):43-6. PMID 25282771
- [Background] Hildenbrand KJ, Vasavada AN. Collegiate and high school athlete neck strength in neutral and rotated postures. J Strength Cond Res. 2013 Nov;27(11):3173-82. doi: 10.1519/JSC.0b013e31828a1fe2. PMID 23439331
- [Background] Daneshvar DH, Riley DO, Nowinski CJ, McKee AC, Stern RA, Cantu RC. Long-term consequences: effects on normal development profile after concussion. Phys Med Rehabil Clin N Am. 2011 Nov;22(4):683-700, ix. doi: 10.1016/j.pmr.2011.08.009. Epub 2011 Sep 23. PMID 22050943
- [Background] Collins CL, Fletcher EN, Fields SK, Kluchurosky L, Rohrkemper MK, Comstock RD, Cantu RC. Neck strength: a protective factor reducing risk for concussion in high school sports. J Prim Prev. 2014 Oct;35(5):309-19. doi: 10.1007/s10935-014-0355-2. PMID 24930131
- [Background] Gutierrez GM, Conte C, Lightbourne K. The relationship between impact force, neck strength, and neurocognitive performance in soccer heading in adolescent females. Pediatr Exerc Sci. 2014 Feb;26(1):33-40. doi: 10.1123/pes.2013-0102. Epub 2013 Oct 2. PMID 24091298

DOCUMENTS (1):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03237468/Prot_000.pdf